CLINICAL TRIAL: NCT02815384
Title: Assessment Of MRI In Patients With Implanted Cardiac Devices
Acronym: MRIPACER
Status: Withdrawn | Type: Observational
Why Stopped: Investigator is leaving the University.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 1605560370
Record Dates: First submitted 2016-05-26; First posted 2016-06-28 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2017-10

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The research goal is to continue to add to the extensive body of peer-reviewed evidence that demonstrates MRI may be safely performed in patients with cIEDs, after they have been evaluated and cleared by cardiology. This study will allow the researchers to collect data from the facilities ongoing clinical practice regarding the number and types of any adverse clinical reactions, and also to document any changes in the implanted cardiac device that may have occurred during the MRI scan. The researchers will also be assessing the results of the MRI and how the imaging findings impact patient care and the clinical outcome of the patient. This data will then be presented to the FDA and the Centers for Medicare and Medicaid Services to further influence federal guidelines and payment structures.

DETAILED DESCRIPTION:
Cardiac implantable electronic devices (cIEDs) generally refer to implanted pacemakers and defibrillators for patients with cardiac disorders affecting their heart rhythm. Previously, cIEDs have been regarded as a contraindication to magnetic resonance imaging (MRI) scans, with concerns that the magnetic fields of the MRI may cause problems with the patient's cIED. However, this is a major healthcare issue, as approximately 50-75% of patients with implanted cIEDs are expected to need a future MRI as part of their clinical care. The inability to get such a test may negatively impact the ability to diagnose and treat future diseases.

However, many of the initial concerns regarding the capability of performing MRI in patients with cIED have likely been overstated. There is peer-reviewed literature dating back to the 1990s regarding the ability to safely perform MRI in patients with cIEDs, if certain protocols are followed regarding patient selection and monitoring. In 2011, Nazarian et al from Johns Hopkins University published a study on 438 patients with cIED that received MRI. There were no adverse clinical effects from this study. In fact, the American College of Radiology updated it's guidance document for Safe MR Practices, and cIEDs are no longer listed as a relative contraindication to obtaining an MRI. However, the presence of cIEDs are still regarded as a relative contraindication to performing MRI at some centers. In addition, performance of MRI in the setting of cIED is denied by the Centers for Medicare and Medicaid Services. Continued accrual of data regarding the safety of performing MRI in patients with cIEDs is needed, including outcomes studies that document the clinical impact of improved diagnostics provided by the MRI on patient care.

ELIGIBILITY:
Inclusion Criteria:

* All patients that require an MRI as part of the normal course of their medical care that also have a cIED and are candidates for MRI .

Exclusion Criteria:

* patient does not require an MRI for their medical care
* patient does not have a cIED
* patient has not been seen or approved by cardiology to be a candidate for MRI
* patients under the age of 18
* pregnant patients
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that require an MRI as part of the normal course of their medical care that also have a cIED and are candidates for MRI .
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Safety of MRI, adverse clinical events | immediately post MRI
  collect safety data

SECONDARY OUTCOMES:
Impact to Patient Care | 6 months
  assess the results of the MRI and how the imaging findings impact patient care
Morbidity, Number of hospitalizations | 6 months
  collected from medical record
Mortality, outcome of death | 6 months
  collected from medical records and phone calls

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Kalb, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center-Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No